CLINICAL TRIAL: NCT06437795
Title: Effectiveness of Dry Needling Versus Cupping Therapy for Pain in Piriformis Syndrome
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Superior University (Other)
Responsible Party: Principal Investigator, Muhammad Naveed Babur, Principal Investigator, Superior University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: MSRSW/Batch-Fall22/715
Record Dates: First submitted 2024-05-25; First posted 2024-05-31 (Actual); Last update posted 2024-05-31 (Actual); Status verified 2024-05

CONDITIONS: Piriformis Syndrome
MeSH Terms: conditions — Piriformis Muscle Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dry Needling Group (Experimental)
  Interventions: Diagnostic Test: Dry Needling Group
- Cupping Therapy Group (Other)
  Interventions: Other: Cupping Therapy Group

INTERVENTIONS:
Diagnostic Test: Dry Needling Group — Participants in this group will receive dry needling therapy. This involves inserting thin needles into trigger points in the piriformis muscle to relieve pain and muscle tension. The therapy will be administered twice a week for 4 weeks, with each session lasting approximately 30 minutes.
  Arms: Dry Needling Group
Other: Cupping Therapy Group — Participants in this group will receive cupping therapy. This involves placing cups on the skin to create suction, which is believed to improve blood flow and reduce muscle tension. The therapy will be administered twice a week for 4 weeks, with each session lasting approximately 30 minutes.
  Arms: Cupping Therapy Group

SUMMARY:
This study aims to compare the effectiveness of two popular therapeutic interventions, dry needling and cupping therapy, in alleviating pain associated with Piriformis Syndrome. Piriformis Syndrome is a neuromuscular disorder caused by the compression or irritation of the sciatic nerve by the piriformis muscle, leading to buttock pain and radiating numbness.

DETAILED DESCRIPTION:
The study will recruit participants diagnosed with Piriformis Syndrome and will randomly assign them to receive either dry needling or cupping therapy over a specific period. The primary outcome will be the reduction in pain intensity measured by standardized pain assessment tools. Secondary outcomes will include improvements in functional mobility and quality of life. By analyzing the efficacy and patient-reported outcomes of both therapies, the study aims to provide evidence-based recommendations for clinicians treating Piriformis Syndrome.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged between 18 to 65 years.
* Diagnosed with piriformis syndrome.
* Experiencing chronic pain for at least 3 months.
* Willingness to comply with the study protocol and attend all therapy sessions.

Exclusion Criteria:

* Recent surgery on the lower back or hip.
* Presence of systemic diseases affecting muscle function (e.g., multiple sclerosis, rheumatoid arthritis).
* Pregnant or breastfeeding women.
* Use of anticoagulant medication or having a bleeding disorder.
* Participating in another clinical trial simultaneously

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2023-11-01 (Actual); Primary Completion 2024-05-01 (Actual); Study Completion 2024-09-01 (Estimated)

PRIMARY OUTCOMES:
Visual Analog Scale (VAS) | 12 Months
  Participants will rate their pain on a scale from 0 (no pain) to 10 (worst possible pain) at the beginning and end of the study.
Oswestry Disability Index (ODI) | 12 months
  This tool assesses the degree of disability in performing daily activities. Quality of life improvements measured by the SF-36 Health Survey, which evaluates physical and mental health status.

CONTACTS AND LOCATIONS:
Locations (1):
- Ghurkee Hospital, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No